CLINICAL TRIAL: NCT05604235
Title: Effectiveness of Oncological Physiotherapy With Neurodynamics and Kinesitherapy (Active+Passive) on Painful Shoulder Cervical Ganglion Post Cervical Evacuation in Head and Neck Cancer Due to Accessory Spinal Nerve of the Accessory Spinal Nerve
Brief Title: Effectiveness of Oncological Physiotherapy on Painful Shoulder Cervical Ganglion in Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHUNSC_2021_91
Record Dates: First submitted 2022-10-27; First posted 2022-11-03 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Shoulder Pain; Rehabilitation
Keywords: cervical lymph node dissection; iatrogenic damage; spinal accessory nerve; physiotherapy
MeSH Terms: conditions — Neoplasms; Shoulder Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic strength exercise group (Experimental): A treatment with therapeutic strength exercises, twice a week, for two months, with a total of 10 exercises, with 20 repetitions each, aimed at improving the strength of the trapezius and sternocleidomastoid muscles mainly, as well as improving mobility in flexion, abduction and rotation of the affected upper limb. The protocol will be carried out in approximately 30 minutes.
  Interventions: Other: Therapeutic upper limb strength exercise treatment
- Passive mobilization group (Experimental): A treatment with passive kinesitherapy, where the physiotherapist will perform the movements of flexion, abduction and rotation of the shoulder, without the patient's intervention; active kinesitherapy, where the patient will perform specifically prescribed movements, without weight, to improve the articular and muscular balance of the scapulohumeral complex and neurodynamics, where mobilisations of the accessory spinal nerve will be performed through therapeutic exercise and manual neurodynamic therapy. This treatment will be carried out once a week for two months in 30-minute sessions.
  Interventions: Other: Treatment with passive and active mobilization of the upper limb.

INTERVENTIONS:
Other: Therapeutic upper limb strength exercise treatment — A treatment with therapeutic strength exercises, twice a week, for two months, with a total of 10 exercises, with 20 repetitions each, aimed at improving the strength of the trapezius and sternocleidomastoid muscles mainly, as well as improving mobility in flexion, abduction and rotation of the affected upper limb. It will take approximately 30 minutes.
  Arms: Therapeutic strength exercise group
Other: Treatment with passive and active mobilization of the upper limb. — A treatment with passive kinesitherapy, where the physiotherapist will perform the movements of flexion, abduction and rotation of the shoulder, without the patient's intervention; active kinesitherapy, where the patient will perform specifically prescribed movements, without weight, to improve the articular and muscular balance of the scapulo-humeral complex and neurodynamics, where mobilizations of the accessory spinal nerve will be performed through therapeutic exercise and manual neurodynamic therapy. This treatment will be carried out once a week for two months in 30-minute sessions.
  Arms: Passive mobilization group

SUMMARY:
Objective: To estimate whether oncological physiotherapy treatment with neurodynamic and kinesitherapy (passive and active) in patients with "painful shoulder due to accessory spinal nerve dissection" operated on for head and neck cancer is more effective than standard therapeutic exercise therapy with strength.

Design: Randomized Clinical Trial (intervention study, no drugs). Two branches of rehabilitative treatment applied by oncological physiotherapist.

GROUP I: Treatment of passive and active mobilizations together with neurodynamics techniques.

GROUP II (or control group) Current treatment applied as gold standard, consisting of therapeutic strength exercise, which the patient will carry out under the supervision of the physiotherapist.

The frequency of both will be twice a week for two months.

Study subjects: Participants who underwent cervical ganglion dissection surgery for head and neck cancer, and who have, as a surgical sequela, a painful shoulder due to accessory spinal nerve injury.

Determinations: At baseline (t0), at one month (t1m) and at the end (t6m) will be measured, (1) the degree of pain of the participants through the pain scale (EVA), (2) the functionality of the shoulder, with the DASH scale and goniometry, (3) the quality of life with the QLQ H&N35 questionnaire, (4) the strength with a hand dynamometer and (5) the degree of neurodynamics of the accessory spinal nerve with the neurodynamic test for this nerve.

DETAILED DESCRIPTION:
Incident cases of painful shoulder due to accessory spinal nerve injury after cervical lymph node dissection in patients with head and neck cancer. Given that clinical data indicate that at least 60% of patients with cervical lymph node dissection have iatrogenic accessory spinal nerve damage, and that the sequelae significantly impair the patient's quality of life, an improvement in quality of life of up to 30% of the QLQ H&N35 score is considered to be significant.

Participants will be selected through the Spanish Association Against Cancer's needs assessment and first impact service, which receives patients from different hospitals. The investigators will make a first appointment with patients likely to be included in the study to check whether they meet the inclusion/exclusion criteria and collect the necessary data.

The investigators will then proceed to randomization to one of the treatment arms. The planned time for the application of the therapy is 2 months. During the course of the clinical trial the participants will attend treatment twice or once a week with a session duration of approximately 30 minutes.

Participants will be seen three times at the oncological physiotherapy service of the AECC during the course of the study [t0, t1 and 6tf]. A first one as mentioned above, an intermediate one after one month and a last one at the end of the clinical trial 2 months after inclusion.

At each of the 3 visits, data on the different variables will be collected: the VAS scale, the QLQ H&N35 quality of life questionnaire and the DASH questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer located in the head and neck.
* Different types of cancer, undergoing cervical lymph node dissection between levels II and V, with pain and/or functional impotence in the shoulder.

Exclusion Criteria:

* Patients with bone metastases
* Patients with functional limitations in the shoulder prior to surgery or that can be demonstrated to be due to other causes.
* Patients who are minors
* Incident cases of painful shoulder in patients with
* Cervical level I lymph node dissection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Eortc QLQ H&N35 questionnaire | Change from baseline at 3 months
  The EORTC Quality of Life questionnaires are developed to assess the quality of life of cancer patients, includes 35 items and scales employ a 4-point response format (''not at all" to ''very much"). A higher score indicates better health

SECONDARY OUTCOMES:
Visual analogue scale | Change from baseline at 3 months
  The visual analogue scale (VAS) is a 10cm long line where 0 indicates no pain at all and 10 the worst pain imaginable. It is a tool that has shown good reliability values (r = 0.94).
The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Change from baseline at 3 months
  It is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale. Scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb
Handgrip strength test | Change from baseline at 3 months
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. Handgrip strength will be measured by handgrip dynamometer (JAMAR). Low grip strength is associated with poor healthcare outcomes and

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Centro Investigación Fisioterapia y Dolor, Alcalá de Henares, Madrid
  - Physiotherapy and Pain Institute, Alcalá de Henares, Madrid
  - Patricia Martinez Merinero, Alcalá de Henares, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Garcia R, Abuin-Porras V, Pecos-Martin D, Romero-Morales C. Effectiveness of Oncological Physiotherapy on Shoulder Dysfunction After Cervical Lymph Node Dissection in Head and Neck Cancer: A Pilot Randomized Controlled Trial. Medicina (Kaunas). 2025 Sep 10;61(9):1636. doi: 10.3390/medicina61091636. PMID 41011027